CLINICAL TRIAL: NCT03945669
Title: Intramedullary Nailing Versus External Ring Fixation for Surgical Treatment of Tibial Shaft Fractures in Adults and Their One Year Outcome on Recovery: Study Protocol for a Pragmatic Randomized Controlled Trial (The IMVEX Trial)
Brief Title: Intramedullary Nailing vs External Ring Fixation for the Treatment of Tibial Shaft Fractures
Acronym: IMVEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Collaborators: Danish Council for Independent Research (Other)
Responsible Party: Principal Investigator, Rasmus Elsøe, Head of Orthopaedic trauma, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LERG1
Record Dates: First submitted 2019-05-03; First posted 2019-05-10 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Tibial Shaft Fracture
Keywords: External ring fixation; Intramedullary nailing; Tibial shaft fracture; patient reported outcome
MeSH Terms: interventions — Fracture Fixation, Intramedullary

STUDY DESIGN:
Intervention Model Description: This study is a multicenter pragmatic assessor blinded randomized and prospective clinical trial.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the study participants, care providers and investigator can not be blinded. The outcome assessor will be blinded with regards to the two treatment groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intramedullary Nail (Active Comparator): Intramedullary Nailing: Alignment will be obtained by closed or limited open reduction of the fracture. A standard reamed intramedullary nail is inserted. Access above the patella, through the patella tendon or parapatellar access is used according to surgeon preferences. One or more cortical screws may be used if deemed appropriate due to fracture pattern. Patients are administered preoperative antibiotics (Dicloxacillin) 15 minutes before surgery commences. Postoperative antibiotics is administered by discretion of the surgeon based on individual patient considerations.
  Interventions: Procedure: Intramedullary Nailing
- External Ring fixator (Experimental): External Ring fixation: Closed or limited open reduction of the fracture is performed. A circular frame is attached on both sides of the fracture. Connection to the bone is obtained by hydroxyapatite coated half pins and/or k-wires with olives as needed according to surgeon preferences. One or more cortical screws may be used if deemed appropriate due to fracture pattern. After applying the ring fixator alignment is assessed radiologically and corrected both peri- and postoperatively. Patients are administered preoperative antibiotics (Dicloxacillin) preoperatively 15 minutes before surgery commences. Following surgery antibiotics are continued until wounds, pin- and wire perforations are dry.
  Interventions: Procedure: External Ring fixation

INTERVENTIONS:
Procedure: Intramedullary Nailing — fracture fixation of the tibial shaft fracture with an intramedullary nail.
  Arms: Intramedullary Nail
Procedure: External Ring fixation — fracture fixation of the tibial shaft fracture with an external ring fixator.
  Arms: External Ring fixator

SUMMARY:
This study is a multicenter pragmatic assessor blinded randomized and prospective clinical trial in which standard intramedullary nailing is compared with external ring fixator for patients with tibial shaft fractures.

DETAILED DESCRIPTION:
This study is a multicenter pragmatic assessor blinded randomized and prospective clinical trial in which standard intramedullary nailing is compared with external ring fixator for patients with tibial shaft fractures.

The primary aim of the project is to compare the one-year Knee Injury and Osteoarthritis Outcome Score - Sport (KOOS-Sport) after standard intramedullary nailing with external ring fixation for patients with tibial shaft fractures.

The explorative aim is to report the effect of the two surgical procedures on the development of complications, time to bone union, pain reactions, muscle strength, activity of daily living and time to return to work.

ELIGIBILITY:
Inclusion Criteria:

* Fracture of the tibial shaft
* OTA classification Type: 42-A1-A3, -B1-B3 and -C1-C3
* The fracture type is deemed operable by intramedullary nail

Exclusion Criteria:

* Below 18 years of age
* Open fracture
* History of severe systemic diseases or cancer
* Bilateral tibial shaft fracture
* Multi fracture patients
* Pregnancy
* Patients without gait function prior to fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
The Knee Injury and Osteoarthritis Outcome Score - sport (KOOS Sport) | 12 month follow up
  KOOS-sport is a standardized and validated patient-reported instrument used in order to assess knee and knee associated problems with regards to activity. The subscale sport is one five subscales: pain, ADL, symptoms, sport and QOL in the KOOS questionnaire . A total score of 100 indicates no symptoms, and 0 indicates major symptoms.

SECONDARY OUTCOMES:
Perceived Pain | 6 weeks, 3+6+12 months
  Development in pain in the two groups will be recorded by patient-reported pain intensity measured on a 10 cm visual analogue scale (VAS) with endpoints "no pain" and "maximal pain" for the worst pain during the last 24 hours and resting pain.
Patient-reported pain reactions | 6 weeks, 3+6+12 months
  Pain DETECT questionnaire. The painDETECT screening questionnaire (PD-Q), uses a scoring method between - 1 and 38 to estimate the likelihood of a neuropathic pain component in patients.
Pain sensitivity | 6 weeks, 3+6+12 months
  Pain sensitivity will be assessed by pressure pain thresholds (PPTs) recorded by handheld pressure algometry (Algometer Type II, Somedic AB, Sweden).
Muscle strength | 6+12 months
  Isometric muscle strength in the two groups will be measured by a strap-mounted dynamometer attached to the wall (Mecmesin AFG2500, Mecmesin Ltd, West Sussex, UK). Girth measures of thigh and calf will be used to examine muscle atrophy and/or effusion
Time to bone union | 6 weeks, 3+6+12 months
  Bone union, in the two surgical groups will be evaluated on standard AP and side X-rays of the fractured leg. The evaluation of bone union will be defined as: i) visible callus formation on at least three of four sides, no visible fracture line and no pain from fracture site at weight-bearing and during clinical examination.
Radiological alignment | 6 weeks, 3+6+12 months
  Alignment of the tibia will be evaluated using the EOS scanning system.
Health related QOL | 6 weeks, 3+6+12 months
  Eq5D-5L is a standardized questionnaire developed to assess general health outcome (29). It consists of five dimensions: Mobility, self-care, usual activities, pain/discomfort and anxiety/depression, and a self-rated health scale on a 20 cm vertical, visual analogue scale with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine'. An Eq5d-5L index of 1.0 indicated full health, 0 death, and -0.59 denoted a condition worse than death
Time to return to work | 6 weeks, 3+6+12 months
  Measure the time from surgery to end of sick leave measured in days.
Health economic evaluation | 12 months
  Measure the cost of treatment in the two groups within the first year following surgery
Gait assessment | 3+6+12 months
  Gait asymmetries will be measured with patients walking on a pressure-sensitive mat.
Patient Acceptable Symptom State (PASS) | 3+6+12 months
  This instrument evaluate when the patient reaches a acceptable patient observed pain and function level, where the patient no longer demands treatment
The Knee Injury and Osteoarthritis Outcome Score (KOOS) | 6 weeks, 3+6+12 months
  KOOS is a standardized and validated patient-reported instrument used in order to assess knee and knee associated problems.The questionnaire includes five subscales: pain, ADL, symptoms, sport and QOL. A total score of 100 indicates no symptoms, and 0 indicates major symptoms.
Foot And Ankle Outcome Score (FAOS) | 6 weeks, 3+6+12 months
  FAOS is a standardized and validated patient-reported instrument used in order to assess foot and ankle associated problems divided into 5 subscales. The questionnaire includes five subscales: pain, ADL, symptoms, sport and QOL. A total score of 100 indicates no symptoms, and 0 indicates major symptoms.

OTHER OUTCOMES:
Adverse events | 6 weeks, 3+6+12 months
  Adverse events, defined as any negative or unwanted reactions to the two surgical procedures, will be recorded. These will include deep infection, pin infection, skin infections, malalignment, compartment syndrome or any other reported physical discomfort. An adverse effects committee will manage adverse reactions at the time of the adverse reaction.

CONTACTS AND LOCATIONS:
Overall Officials: Rasmus Elsøe, PhD, Study Director — Aalborg University Hospital; Rasmus Stokholm, MD, Principal Investigator — Aalborg University Hospital; Peter Larsen, PhD, Principal Investigator — Aalborg University Hospital
Locations (3):
- Denmark (3):
  - Aalborg University Hospital, Department of orthopaedic surgery, Aalborg
  - Aarhus University Hospital, Aarhus
  - Regional Hospital Viborg, Viborg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Larsen P, Stokholm R, Rolfing JD, Petruskevicius J, Rasmussen MK, Jensen SS, Elsoe R. Intramedullary nailing versus external ring fixation for tibial shaft fractures: an explorative analysis of muscle strength from the IMVEX trial. Arch Orthop Trauma Surg. 2025 Jul 18;145(1):379. doi: 10.1007/s00402-025-05995-6. PMID 40679543